CLINICAL TRIAL: NCT01136265
Title: Dual-time PET/CT and Sentinel Node Diagnostics Preoperatively in Patients With Oral Cancer
Brief Title: PET/CT and Sentinel Node in Oral Cancer
Acronym: PETNode
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Dr. Christine Winkler Duemcke, Dep. of Nuclear Medicine & PET, Rigshospitalet
Other Study IDs: RH-238_10
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-06

CONDITIONS: Oral Cancer
Keywords: dual-time PET/CT; sentinel node
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, primary cancer tissue, normal oral tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators want to pre-operatively scan patients who do not have any clinically suspicion of metastases with an 18F-FDG-PET/CT whole body scan , where after they go to lymphoscintigraphy incl. SPECT/CT and sentinel node biopsy. Material from the oral cancer and, after permission of each patient, also normal oral tissue will be analyzed molecular-biologically. Also a blood sample will be analyzed for molecular tumor markers.

The investigators want to see if PET/CT is able to detect any signs of sub-clinically metastases. Besides, the investigators want to fusion PET/CT with SPECT/CT data from the lymphoscintigraphy study and improve our PET/CT scanning with a dual-time PET scan of the head-and-neck region.

DETAILED DESCRIPTION:
These patients are normally preoperatively sent to a CT scan of the thorax and abdomen; in this study, this CT is replaced by a wholebody PET/CT scan. Afterwards, the patients goes to sentinel node lymphoscintigraphy and then to operation.

By combining biomarkers and molecular imaging in patients with a clinically T1/T2N0M0 oral cancer, we want to characterize the tumor physiologically and correlate these physiological features to the clinical appearance of the cancer.

Aims of the study:

* can PET/CT in this patient group metastases with consequently change of treatment?
* can fusion of SPECT/CT and PET/CT with calculation of standardized uptake value (SUV) indicate, how much tumor tissue there should be in a positive sentinel node to be detected by PET?
* can dual-time PET scanning better determine lymph node metastases, than single-time PET scanning?
* correlation between SUV in PET with molecular-biological findings both in the primary tumor and in metastases

ELIGIBILITY:
Inclusion Criteria:

* biopsy-verified oral cancer
* over 18 years of age

Exclusion Criteria:

* under 18 years of age
* inable patients
* pregnancy
* known allergy to contrast agents
* kidney insufficiency
* other known cancer
* diabetes mellitus
* acute medical conditions such as acute infection, acute cardial or lung disease or other intercurrent diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 consecutive patients with biopsy-verified oral cancer without a suspicion of metastases and without prior treated neck
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine W Dümcke, Dr., Principal Investigator — Dep. of Nuclear Medicine & PET
Locations (2):
- Denmark (2):
  - Dep. of Nuclear Medicine & PET, Copenhagen
  - Dep. of otorhinolaryngology, Head & Neck Surgery/ Rigshospitalet, Copenhagen